CLINICAL TRIAL: NCT00464282
Title: Fluorine-18-α-Methyltyrosine Positron Emission Tomography for Diagnosis and Staging of Lung Cancer
Status: Completed | Type: Observational
Sponsor: Gunma University (Other)
Other Study IDs: Gunma 444
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Fluorine-18-α-methyltyrosine,; Positron emission tomography,; Fluorodeoxyglucose; Lung cancer,; Amino acid transportor 1,; Ki-67; Proven or suspected non-small cell lung cancer were enrolled in the study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Objective: L-[3-18F]-α-methyltyrosine (FMT) is an amino-acid tracer for PET. We evaluated the diagnostic usefulness of 18F-FMT PET in non-small cell lung cancer (NSCLC) patients. Tumor uptake of 18F-FMT PET was compared with 18F-FDG PET and the correlation with L-type amino acid transporter 1 (LAT1) expression also investigated.

Method: Fifty patients with NSCLC were enrolled in this study, and a pair of PET study with 18F-FMT and 18F-FDG was performed. LAT1 expression and Ki-67 labeling index of the resected tumors were analyzed by immunohistochemical study.

ELIGIBILITY:
Inclusion Criteria:

* proven or suspected non-small cell lung cancer

Exclusion Criteria:

* uncontrolled diabetes mellitus

Ages: 8 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: kyoichi kaira, MD, Principal Investigator — Gunma Unversity Graduate School of Medicine

REFERENCES:
- [Derived] Kaira K, Oriuchi N, Shimizu K, Tominaga H, Yanagitani N, Sunaga N, Ishizuka T, Kanai Y, Mori M, Endo K. 18F-FMT uptake seen within primary cancer on PET helps predict outcome of non-small cell lung cancer. J Nucl Med. 2009 Nov;50(11):1770-6. doi: 10.2967/jnumed.109.066837. Epub 2009 Oct 16. PMID 19837768